CLINICAL TRIAL: NCT03873818
Title: A Phase II Study of Open Label Low Dose Ipilimumab in Combination With Pembrolizumab in Metastatic Melanoma Patients With Brain Metastases
Brief Title: Low Dose Ipilimumab With Pembrolizumab in Treating Patients With Melanoma That Has Spread to the Brain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0875; NCI-2019-00406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0875 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-19; First posted 2019-03-13 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8
MeSH Terms: conditions — Brain Neoplasms; Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ipilimumab, pembrolizumab) (Experimental): Patients receive ipilimumab IV over 90 minutes and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 4 cycles for ipilimumab and up to 35 cycles for pembrolizumab in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies the side effects and how well low dose ipilimumab works in combination with pembrolizumab in treating patients with melanoma that has spread to the brain. Immunotherapy with monoclonal antibodies, such as ipilimumab and pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess clinical benefit rate (CBR), defined as complete response (CR) + partial response (PR) + stable disease (SD) > 6 months, in the brain in subjects with melanoma brain metastasis (MBM) per modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria who are treatment naive to anti-PD-1 agents in the metastatic setting (prior adjuvant anti-PD1 allowed).

SECONDARY OBJECTIVES:

I. To assess clinical benefit rate (CBR) in the brain in subjects with MBM per modified RECIST 1.1 in patients who previously progressed on PD-1 inhibitors.

II. To assess overall survival (OS) and progression free survival (PFS). III. To evaluate the brain-specific safety and tolerability of the combination regimen in subjects with or without stereotactic radiotherapy (SRT) received prior to study entry, or on study.

IV. To evaluate cytokine levels and changes in the T-cell population in the cerebrospinal fluid (CSF) and blood in patients treated with combination low dose ipilimumab and pembrolizumab.

V. To assess changes in relative apparent diffusion coefficient as measured by magnetic resonance imaging (MRI) as an early predictor of response.

VI. To assess changes in circulating cfDNA (cell-free deoxyribonucleic acid) as determinants of response and/or markers of early progression.

VII. To evaluate molecular and immunological changes in extracranial lesions.

OUTLINE:

Patients receive ipilimumab intravenously (IV) over 90 minutes and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 4 cycles for ipilimumab and up to 35 cycles for pembrolizumab in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 6 weeks for the first year, and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 12 weeks.
* Subjects must have signed and dated an IRB/IEC (Institutional Review Board/Independent Ethics Committee) approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
* Histologically confirmed malignant melanoma with measurable metastases in the brain (>= 0.5 cm).
* At least one measurable intracranial target lesion, which previously was not treated with local therapy (no prior stereotactic radiosurgery [SRS] to this lesion). Largest diameter of >= 0.5 cm, but =< 3 cm as determined by contrast-enhanced MRI.
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks are preferred) OR at least 4 unstained slides with an associated pathology report for testing of tumor PD-L1 expression:

  * Tumor tissue should be of good quality based on total and viable tumor content.
  * Patients who do not have tissue specimens may undergo a biopsy during the screening period. Acceptable samples include core-needle biopsies for deep tumor tissue or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions.
  * Tumor tissue from bone metastases is not evaluable for PD-L1 expression and is therefore not acceptable.
  * However, if repeat biopsy is not feasible, and no archival tissue available patient still may be enrolled
* Prior stereotactic radiotherapy (SRT) and prior excision of up to 5 MBM is permitted if there has been complete recovery, with no neurologic sequelae, and measurable lesions remain. Growth or change in a lesion previously irradiated will not be considered measurable. Regrowth in cavity of previously excised lesion will not be considered measurable. Note: Any prior SRT to brain lesions or prior excision must have occurred >= 2 weeks before the start of dosing for this study.
* Prior radiation to non-central nervous system (non-CNS) is allowed, and does not require a washout period for treatment initiation.
* Subjects must be free of neurologic signs and symptoms related to metastatic brain lesions and must not have required or received systemic corticosteroid therapy in the 10 days prior to beginning protocol therapy.
* ECOG (Eastern Cooperative Oncology Group) performance status =< 1.
* Absolute neutrophil count >= 1500/uL.
* Platelets >= 100,000/uL.
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L.
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 30 L/min with creatinine levels > 1.5 x institutional ULN. GFR (glomerular filtration rate) can also be used in place of creatinine or CrCl (creatinine clearance).
* Total bilirubin =< 1.5 ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases).
* International normalized ratio (INR) OR prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Women of child-bearing potential (WOCBP) must not be breastfeeding and must have a negative pregnancy test within 3 days prior to initiation of dosing. She must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 120 days after the last dose of study drug. WOCBP must agree to adhere to the contraceptive guidance in the protocol. Note: A female participant is eligible to participate if she is not a woman of childbearing potential as defined by the protocol.
* Fertile men must agree to use an acceptable method of birth control as described in the protocol while on study drug and up to 120 days after the last dose of study drug and also refrain from donating sperm during this period.
* All associated toxicity from previous or concurrent cancer therapy must be resolved (to =< grade 1 or baseline) prior to study treatment administration.
* Steroids for physiological replacement are allowed.

Exclusion Criteria:

* History of known leptomeningeal involvement (lumbar puncture not required).
* Previous stereotactic or highly conformal radiotherapy within 2 weeks before the start of dosing for this study. Note the stereotactic radiotherapy field must not have included the brain index lesion(s).
* Subjects previously treated with SRT > 5 lesions in the brain
* Brain lesion size > 3 cm.
* Prior checkpoint inhibitor therapy. Allowable prior therapy: Approved adjuvant therapies, which may include molecularly-targeted agents, IFN-·, and ipilimumab.

  * Patients who received ipilimumab as adjuvant or neoadjuvant therapy must have a 6 month washout before receiving any dosing on this study.
  * Cohort A: Prior anti-PD in the adjuvant setting is allowed, but washout period is 6 months.
  * For Cohort B: Patients with unresectable metastatic melanoma who received either anti-PD-1 or PDL-1 in the past are eligible. Washout period a minimum 3 weeks.
* Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with major medical, neurologic or psychiatric condition who are judged as unable to fully comply with study therapy or assessments should not be enrolled.
* Subject has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. Note: The time requirement does not apply to participants who underwent successful treatment of superficial bladder cancer, in situ cervical cancer, or other in-situ cancers. Subjects with a completely treated prior malignancy and no evidence of disease for >= 2 years are eligible.

  * Skin cancer exclusion: Please note that basal cell carcinoma and squamous cell carcinoma is exempt from needing resection prior to treatment. (Resection can be completed after the start of treatment).
* Has a known history of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (hepatitis C virus [HCV] ribonucleic acid (RNA) [qualitative] is detected). Note: Without known history, testing needs to be performed to determine eligibility. Hepatitis C antibody (Ab) testing is allowed for screening purposes in countries where HCV RNA is not part of standard of care.
* Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
* The use of corticosteroids is not allowed for 10 days prior to initiation of therapy (based upon 5 times the expected half-life of dexamethasone) except patients who are taking steroids for physiological replacement. If alternative corticosteroid therapy has been used, consultation with the sponsor medical monitor is required to determine the washout period prior to initiating study treatment.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study initiation. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Subjects with history of life-threatening toxicity related to prior ipilimumab adjuvant therapy except those that are unlikely to re-occur with standard countermeasures (e.g. hormone replacement after adrenal crisis).
* Major surgical procedure, open biopsy (excluding skin cancer resection), or significant traumatic injury within 14 days of initiating study drug (unless the wound has healed) or anticipation of the need for major surgery during the study.
* Non-healing wound, ulcer, or bone fracture.
* Women who are breast-feeding or pregnant.
* Uncontrolled intercurrent illness (i.e., active infection >= grade 2) or concurrent condition that, in the opinion of the Investigator, would interfere with the study endpoints or the subject's ability to participate.
* History of clinically significant cardiac disease or congestive heart failure > New York Heart Association (NYHA) class 2. Subjects must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months.
* Investigational drug use within 14 days (or 5 half-lives, whichever is longer) of the first dose of ipilimumab and pembrolizumab.
* Has a history of non-infectious pneumonitis that required steroids or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabella C Glitza, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Low Dose Ipilimumab in Combination with Pembrolizumab in Metastatic Melanoma patients with brain metastases
Groups:
- Cohort A: Treatment Naïve; Cohort B: Previously Progressed on PD-1 Inhibitors: Ipilimumab 1 mg/kg IV q3 wks (up to 4 doses) & Pembrolizumab 200 mg IV q3 wks (up to 35 doses)
Period: Overall Study
Arm/Group | Cohort A: Treatment Naïve | Cohort B: Previously Progressed on PD-1 Inhibitors
Started | 20 | 4
Completed | 10 | 1
Not Completed | 10 | 3
Not completed — Death | 9 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Treatment Naïve | Cohort B: Previously Progressed on PD-1 Inhibitors | Total
Number analyzed (Participants) | 20 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 1 | 11
  >=65 years | 10 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 9
  Male | 11 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 4 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 4 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) in PD-1 naïve Patients
Description: clinical benefit rate (CBR), defined as CR + PR + SD > 6 months, in the brain in subjects with MBM per modified RECIST 1.1 criteria who are treatment naïve to anti-PD-1 agents in metastatic setting (prior adjuvant anti-PD1 allowed).
Time Frame: Baseline to 2 years
Population: For Cohort B- as these patients were not PD-1 naïve, there is no data to be entered in this section. The CBR for this cohort is listed under Secondary outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Treatment Naïve | Cohort B: Previously Progressed on PD-1 Inhibitors
Number analyzed (Participants) | 20 | 0
percentage of participants | 68.4 |

2. Secondary Outcome: CBR for Patients Who Progressed on PD-1 Inhibitors
Description: Assess CBR in the brain in subjects with MBM per modified RECIST 1.1 in patients who previously progressed on PD-1 inhibitors.
Time Frame: Baseline to 2 years
Population: This metric only applies to Cohort B, as this objective only looks ONLY at the patients who are PD-1 refractory (Cohort B by definition)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Treatment Naïve | Cohort B: Previously Progressed on PD-1 Inhibitors
Number analyzed (Participants) | 0 | 4
Participants |  | 1

3. Secondary Outcome: Overall Survival (OS) & Progression-free Survival (PFS)
Description: Assess OS and PFS.
Time Frame: Baseline to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Treatment Naïve | Cohort B: Previously Progressed on PD-1 Inhibitors
Number analyzed (Participants) | 20 | 4
months
  PFS | 11.8 [1.4 to NA] — The upper 95% CI is not estimated due to insufficient number of participants with events. | 1.4 [1.3 to NA] — The upper 95% CI is not estimated due to insufficient number of participants with events.
  OS | NA [5.7 to NA] — Median OS not reached due to insufficient number of participants with events. | 11.0 [8.8 to NA] — The upper 95% CI is not estimated due to insufficient number of participants with events.

4. Secondary Outcome: Brain-specific Safety and Tolerability
Description: Evaluate the brain-specific safety and tolerability of the combination regimen in subjects with or without SRT received prior to study entry, or on study.
Time Frame: Baseline to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Treatment Naïve | Cohort B: Previously Progressed on PD-1 Inhibitors
Number analyzed (Participants) | 20 | 4
Participants
  CNS concerns | 0 | 0
  Treatment related grade 3 or 4 AEs | 5 | 0

ADVERSE EVENTS:
Time Frame: Approximately 4 years and 10 months
Arm/Group | Cohort A: Treatment Naïve | Cohort B: Previously Progressed on PD-1 Inhibitors
All-Cause Mortality (participants affected / at risk) | 9/20 | 3/4
Serious Adverse Events (participants affected / at risk) | 10/20 | 1/4
Other Adverse Events (participants affected / at risk) | 20/20 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Treatment Naïve (N=20) | Cohort B: Previously Progressed on PD-1 Inhibitors (N=4)
Fall (General disorders) | 1 (1) | 0 (0)
Cough/dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (1)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ALT increased (Investigations) | 2 (2) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decrased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Nervous system disorders - Other, left sided hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Treatment Naïve (N=20) | Cohort B: Previously Progressed on PD-1 Inhibitors (N=4)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (19) | 2 (2)
Alkaline phosphatase increased (Investigations) | 6 (8) | 2 (2)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 8 (12) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (18) | 2 (2)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bladder Infection (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Blood and lymphatic system disorders) | 2 (3) | 1 (2)
Blurred vision (Eye disorders) | 4 (4) | 1 (1)
Brusing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1)
Cholesterol High (Investigations) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 6 (6) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Creatinine increased (Investigations) | 9 (15) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (13) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Edema limbs (General disorders) | 4 (4) | 2 (2)
Encephalopathy (Endocrine disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 13 (25) | 3 (4)
Fever (General disorders) | 1 (1) | 1 (1)
Flashing lights (Eye disorders) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 5 (5) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Metabolism and nutrition disorders) | 9 (14) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (11) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (11) | 4 (4)
Hyperkalemia (Investigations) | 2 (2) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 4 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalmeia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 4 (4) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Joint rang of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Left sided hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (13) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 7 (8) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (13) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (9) | 3 (4)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (2) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (2) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Weight loss (Investigations) | 4 (4) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 4 (4) | 0 (0)
Left ear hearing changes (Ear and labyrinth disorders) | 1 (1) | 0 (0)
T4 increased (Endocrine disorders) | 1 (1) | 0 (0)
T4 decreased (Endocrine disorders) | 2 (2) | 0 (0)
T3 decreased (Endocrine disorders) | 2 (2) | 0 (0)
Halo effect aroung light (Eye disorders) | 1 (1) | 0 (0)
Visual disturbance (Eye disorders) | 2 (2) | 0 (0)
Loss of vision- rt side (Eye disorders) | 1 (1) | 0 (0)
COVID (Infections and infestations) | 1 (1) | 0 (0)
Autonomic Dystunction (Immune system disorders) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
WBC elevated (Investigations) | 2 (3) | 0 (0)
Hyperphosphatemia (Investigations) | 2 (2) | 0 (0)
ANC increased (Investigations) | 1 (1) | 0 (0)
T4 increased (Investigations) | 1 (2) | 0 (0)
Urination Hesitation (Renal and urinary disorders) | 1 (1) | 0 (0)
Lesion scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lesion face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Perioral erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen Planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Perleche (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
TSH elevated (mildly) (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03873818/Prot_SAP_000.pdf